CLINICAL TRIAL: NCT01405885
Title: Phase I, Open Label Study to Evaluate Safety, Tolerability and Immunogenicity of Multiple Combinations of H1 and H5 Influenza Hemagglutinin Plasmids Administered ID Followed by in Vivo Electroporation With CELLECTRA®-3P in Healthy Adults
Brief Title: A Study of DNA Vaccine With Electroporation for the Prevention of Disease Caused by H1 and H5 Influenza Virus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Inovio Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FLU-101
Record Dates: First submitted 2011-07-27; First posted 2011-07-29 (Estimated); Last update posted 2014-03-03 (Estimated); Status verified 2014-02

CONDITIONS: Healthy
Keywords: Universal Influenza; Intradermal DNA vaccine; Electroporation; H1 and H5; DNA Vaccination; Influenza; INO-3510
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (10):
- Arm A - 0.9mg of INO-3605 (Experimental)
  Interventions: Biological: INO-3605
- Arm B - 0.9mg of INO-3609 (Experimental)
  Interventions: Biological: INO-3609
- Arm C- 0.9mg of INO-3401 (Experimental)
  Interventions: Biological: INO-3401
- Arm D- 0.3mg of INO-3609 (Experimental)
  Interventions: Biological: INO-3609
- Arm E - 0.45mg each INO-3605 , INO-3609 (Experimental)
  Interventions: Biological: INO-3605 AND INO-3609
- Arm F - 0.3mg each of INO-3401,INO-3605,INO-3609 (Experimental)
  Interventions: Biological: INO-3510
- Arm G - 0.9mg of INO-3609 (Experimental)
  Interventions: Biological: INO-3609
- Arm H - 0.9mg of INO-3609 (Experimental)
  Interventions: Biological: INO-3609
- Arm I - Seasonal influenza vaccine (Active Comparator)
  Interventions: Biological: Seasonal Influenza vaccine
- Arm J - 1.8mg of INO-3609 (Experimental)
  Interventions: Biological: INO-3609

INTERVENTIONS:
Biological: INO-3605 — 0.9mg of INO-3605 vaccine delivered ID followed by electroporation on Day 0, Week 8 and 24.
  Arms: Arm A - 0.9mg of INO-3605
Biological: INO-3609 — 0.9mg of INO-3609 vaccine delivered ID followed by electroporation on Day 0, Week 8 and 24.
  Arms: Arm B - 0.9mg of INO-3609
Biological: INO-3401 — 0.9mg of 3401 vaccine delivered ID followed by electroporation on Day 0, Week 8 and 24.
  Arms: Arm C- 0.9mg of INO-3401
Biological: INO-3609 — 0.3mg of INO-3609 vaccine delivered ID followed by electroporation on Day 0, Week 8 and 24.
  Arms: Arm D- 0.3mg of INO-3609
Biological: INO-3605 AND INO-3609 — 0.45mg each of INO-3605 AND INO-3609 vaccine delivered ID followed by electroporation on Day 0, Week 8 and 24.
  Arms: Arm E - 0.45mg each INO-3605 , INO-3609
Biological: INO-3510 — 0.3mg each of INO-3605, INO-3609 AND INO-3401 vaccine delivered ID followed by electroporation on Day 0, Week 8 and 24.
  Arms: Arm F - 0.3mg each of INO-3401,INO-3605,INO-3609
Biological: INO-3609 — 0.9mg of INO-3609 vaccine delivered ID followed by electroporation on Day 0, Week 16 and 24.
  Arms: Arm G - 0.9mg of INO-3609
Biological: INO-3609 — 0.9mg of INO-3609 vaccine delivered ID followed by electroporation on Day 0 and Week 8
  Arms: Arm H - 0.9mg of INO-3609
Biological: Seasonal Influenza vaccine — 0.5ml of vaccine delivered IM
  Arms: Arm I - Seasonal influenza vaccine
Biological: INO-3609 — 1.8mg of INO-3609 vaccine delivered ID followed by electroporation on Day 0, Week 8 and 24.
  Arms: Arm J - 1.8mg of INO-3609

SUMMARY:
This is a Phase I, parallel design open label study to evaluate safety, tolerability and immunogenicity of nine different formulation of two individual H1 and one H5 HA plasmid administered intradermally followed by electroporation in healthy adults

DETAILED DESCRIPTION:
The use of DNA plasmids containing genes that express viral antigens may be a promising way to formulate a vaccine that can effectively prevent infection and disease caused by the H5N1 avian influenza virus and H1N1 influenza viruses. Plasmid vectors are simple to construct and are easy to manufacture at a relatively low cost. Vaccination with plasmids that express influenza proteins should induce the development of serum antibodies and might also induce significant quantities of secretory IgA antibodies and/or CMI. The DNA sequences included in the vaccine could also result in the proliferation of T lymphocytes that could broaden the effectiveness of the vaccine to include variant strains of H5N1 and H1N1 with antigenically modified HA (i.e., drifted strains).

Electroporation (EP) is a technology in which a transmembrane electrical field is applied to increase the permeability of cell membranes to create microscopic pathways (pores) and thereby enhance the uptake of drugs, vaccines, or other agents into target cells. Their presence allows macromolecules, ions, and water to pass from one side of the membrane to the other. The presence of a constant field influences the kinetics of directional translocation of the macromolecular plasmid, such that the plasmid delivery in vivo has been sufficient to achieve physiological levels of secreted proteins. ID injection of a plasmid followed by EP has been used very successfully to deliver therapeutic genes that encode for a variety of hormones, cytokines, or enzymes in a variety of species. EP is currently being used in humans to deliver cancer vaccines and therapeutics as well as in gene therapy. The expression levels are increased by as much as 3 orders of magnitude over plasmid injection alone.

The use of EP via the CELLECTRA® device should increase the expression of H5N1 and H1N1 influenza virus genes in the study vaccines.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent in accordance with institutional guidelines. If required by local law, candidates must also authorize the release and use of protected health information (PHI);
* Adults of either gender 18-55 years of age at entry;
* Healthy subjects as judged by the Investigator based on medical history, physical examination, and normal results for an ECG, CBC, serum chemistries, and urinalysis done up to 4 weeks prior to enrollment and administration of vaccination ± EP;
* Current nonsmoker;
* Women of child-bearing potential (WOCBP) agree to remain sexually abstinent, use medically effective contraception (oral contraception, barrier methods, spermicide, etc), or have a partner who is sterile (i.e., vasectomy) until 12 weeks after last vaccination;
* Able and willing to comply with all study procedures.

Exclusion Criteria:

* Positive serological test for Human Immunodeficiency Virus, hepatitis C virus or hepatitis B virus surface antigen (HBsAg) or Grade 3 or greater CPK at screening;
* Pregnant or breastfeeding subjects;
* Any concurrent condition requiring the continued use of systemic or topical steroids at or near the injection site (excluding inhaled and eye drop-containing corticosteroids) or the use of other immunosuppressive agents. All other corticosteroids must be discontinued > 4 weeks prior to Day 0 of study vaccine administration;
* Administration of any blood product within 3 months of enrollment;
* Prior receipt of any investigational or licensed H5N1 influenza vaccine at any time;
* Subjects with contraindications to influenza vaccination other than egg allergy (such as a history of Guillain-Barre Syndrome after receiving influenza vaccine);
* Administration of any vaccine within 6 weeks of enrollment;
* Participation in a study with an investigational compound or device within 4 weeks of signing informed consent;
* Subjects with cardiac pre-excitation syndromes (such as Wolff-Parkinson-White);
* Subjects with a history of seizures (unless seizure free for 5 years);
* Subjects with tattoos, scars, or active lesions/rashes within 2 cm of the site of vaccination ± EP;
* Subjects with any implantable leads;
* Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements;
* Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (i.e. infections disease) illness must not be enrolled into this study;
* Any other conditions judged by the investigator that would limit the evaluation of a subject.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 116 (Actual)
Dates: Start 2011-05; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of nine different formulation of multiple combination of H1 and H5 HA plasmid administered ID followed by electroporation in healthy adult subjects | Day 0 through Month 12
  Frequency and severity of local and systemic reactogenicity signs and symptoms, adverse events and serious adverse events

SECONDARY OUTCOMES:
Humoral and cellular immune responses | Day 0 through Month 12
  Magnitude and frequency of antibody and cell mediated immune response to influenza proteins
tolerability and immunogenicity of multiple formulations of H1 and H5 HA plasmids administered ID followed by electroporation to seasonal influenza vaccine | Day 0 through Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Mark Bagarazzi, M.D., Study Director — Inovio Pharmaceuticals
Locations (3):
- United States (3):
  - Miami Research Associates, Miami, Florida
  - Vince and Associates, Overland Park, Kansas
  - SNBL, Baltimore, Maryland

REFERENCES:
- See also: Sponsor's address — http://www.inovio.com